CLINICAL TRIAL: NCT05964140
Title: Should we Use Post-operative Antibiotics Following Surgery for Patients With Mandible Fractures? The MANTRA Trial (MANdibular TRauma and Antibiotic Use)
Brief Title: The MANTRA Trial (MANdibular TRauma and Antibiotic Use)
Acronym: MANTRA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: East Lancashire Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEV008
Record Dates: First submitted 2023-07-11; First posted 2023-07-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mandible Fracture; Post-operative Antibiotics
Keywords: Mandible fractures; Antibiotics; Open Reduction and Internal Fixation; Co-amoxiclav; Antibiotic Resistance; Surgical Site Infection
MeSH Terms: conditions — Mandibular Fractures; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Non-inferiority RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group A: One induction IV dose
  Interventions: Drug: Different post-operative antibiotic regimens following surgical treatment of mandible fractures
- Group B (Experimental): Group B: One induction IV dose and 2 further postoperative IV doses
  Interventions: Drug: Different post-operative antibiotic regimens following surgical treatment of mandible fractures
- Group C (Active Comparator): Group C: One IV dose of antibiotics on induction and 2 further postoperative IV doses (as above), followed by a 5-day course of oral co-amoxiclav 625mg every 8 hours if no penicillin allergy
  Interventions: Drug: Different post-operative antibiotic regimens following surgical treatment of mandible fractures

INTERVENTIONS:
Drug: Different post-operative antibiotic regimens following surgical treatment of mandible fractures — The 3 study arms represent the most common antibiotic regimens used in current clinical practice following surgery for mandible fractures. The control group is the most common approach.
  All patients will receive 1 dose of IV antibiotics (co-amoxiclav 1.2g), if no penicillin allergy, on induction of anaesthesia, prior to their surgery.
  The participants will be randomised to the following (1:1:1):
  Group A: No further antibiotics Group B: 2 further postoperative IV doses of co-amoxiclav 1.2g Group C: 2 further postoperative IV doses (as above), followed by a 5-day course of oral co-amoxiclav 625mg every 8 hours if no penicillin allergy (Control).

SUMMARY:
1. FULL TITLE OF THE PROJECT Should we use post-operative antibiotics following surgery for patients with mandible fractures? The MANTRA trial (MANdibular TRauma and Antibiotic use)
2. SUMMARY OF RESEARCH (ABSTRACT) Research Question: Are post-operative antibiotics required following surgery for patients with mandible fractures? Background: Mandible fractures are the commonest facial fractures needing surgery and account for a significant percentage of the acute workload in Oral & Maxillofacial Surgery (OMFS) units. The UK records over 6000 new cases per year. Patients having surgery for mandible fractures have a theoretical risk of developing surgical site infection, due to the proximity of the fracture lines to the oral cavity microbes and the presence of foreign body (titanium fixation miniplates). For this reason, clinicians often prescribe antibiotics after surgery, to reduce the risk of infection. Previous systematic reviews and a multicentre cohort study performed by this team, revealed significant clinical variation in post-operative antibiotic prescription amongst UK OMFS clinicians and the presence of clinical equipoise. Antibiotic overuse can lead to antibiotic resistance and other antibiotic-related side effects; judicious antibiotic use and stewardship is of paramount importance.

Aim: To determine whether post-operative antibiotics are required at all, following surgery for mandible fractures, and, if so, what is the most clinically- and cost-effective regimen

Objectives:

Primary Objective To conduct a Randomized Controlled Trial (MANTRA) in order to establish the non-inferiority (or not) of not giving post-operative antibiotics versus 2 other post-operative antibiotic regimens. An internal pilot phase will optimise recruitment and retention.

Secondary Objectives

* Measure the cost-effectiveness of the proposed antibiotic pathways
* Assess patient and clinician acceptability to change clinical practice
* Process evaluation to inform dissemination and implementation Methods: The investigators designed and propose the MANTRA RCT to compare 3 post-operative antibiotic approaches to prevent Surgical Site Infections (SSIs) following surgery for mandible fractures. The MANTRA trial is a large open label, multicentre study in NHS OMFS units. The 3 study arms represent the most common clinical pathways in the UK based on previous work; the control group is the approach prescribed by most UK OMFS clinicians. All patients will receive 1 dose of IV antibiotics (co-amoxiclav 1.2g, if no penicillin allergy, which is the most commonly used prophylactic antibiotic currently) on induction of anaesthesia, prior to their surgery.

The participants will be randomised to the following (1:1:1):

Group A: No further antibiotics Group B: 2 further postoperative IV doses of co-amoxiclav 1.2g Group C: 2 further postoperative IV doses (as above), followed by a 5-day course of oral co-amoxiclav 625mg every 8 hours if no penicillin allergy (Control).

Trial processes will be optimised by an internal pilot phase ensuring we recruit, randomise, and retain participants with clear progression criteria. We will also conduct cost-effectiveness analyses and process evaluation for dissemination and implementation

Timeline:

Start of grant: 1st July 2023 Start of RCT / pilot: 1st January 2024 End of pilot: 30th June 2024 End of recruitment: 31st December 2026 End of follow-up: 30th June 2027 Completion: 31st December 2027

Impact and dissemination:

* Practice changing outputs that standardise the use of antibiotics in mandible fractures in the NHS and provide a framework for other surgical prophylaxis research
* A bespoke clinical dissemination plan via an engagement and training legacy
* Cost-effectiveness data to inform policy making
* A research legacy and change of culture in the specialty of OMFS

ELIGIBILITY:
All adult patients aged 18 years or over with mandible fractures requiring surgery. Most of these patients will be identified from the A&E department via the on-call OMFS team or seen in dedicated OMFS trauma clinics. A small proportion of our study population will be seen in an OMFS clinic following referral from GP/GDP.

Inclusion Criteria:

* Ability to provide written informed consent
* Age≥18 years
* Hospital episode of mandible fracture(s)
* Planned treatment is surgery - (ORIF with titanium miniplates)

Exclusion Criteria:

* Isolated mandibular condylar fractures
* Existing fracture site infection
* Immunocompromised (transplant patients, haematological malignancies, HIV/AIDS) - a clear definition will be provided in the protocol
* Pathological fracture (e.g., malignancy, osteoradionecrosis, cysts, Medication-Related Osteonecrosis of the Jaws [MRONJ])
* Fractures open to skin
* Inability to provide written informed consent
* Other injuries or infections mandating ongoing post-operative antibiotics (e.g., panfacial fractures with mandible fracture component)
* Patients allergic to first and second-line antibiotic prophylaxis (as outlined above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2841 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 30 days
  Incidence of Surgical Site Infection (CDC definition) following surgery for mandible fractures

SECONDARY OUTCOMES:
Return to theatre within 30 days | 30 days
Length of hospital stay | 14 days, 30 days, 180 days
Death and cause of death | 14 days, 30 days, 180 days
Hospital readmission | 30 days
Malunion: fracture non-healing | 180 days
  Fibrous union, fracture mobility, absence of callus formation
Malocclusion: teeth not meeting as they should | 180 days
  When the fracture reduction failed to restore the dental occlusion
Metalwork removal | 14 days, 30 days, 180 days
  When the fixation titanium miniplates need to be removed at any point and for any reason
Overall antibiotic exposure | 14 days, 30 days, 180 days
Antibiotic related adverse events/serious adverse events | 14 days, 30 days, 180 days
Cost | 14 days, 30 days, 180 days
HRQoL (EQ-5D-5L) | 14 days, 30 days, 180 days
  Health Related Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Kyzas, PhD, Principal Investigator — Consultant OMFS H&N Surgeon ELHT
Locations (1):
- East Lancashire Hospitals NHS Trust, Blackburn, Lancashire, United Kingdom